CLINICAL TRIAL: NCT02845453
Title: A Randomized Controlled Trial of Quetiapine for the Treatment of Youth With Co-occurring Substance Use Disorders and Severe Mood Dysregulation
Brief Title: Treatment With Quetiapine for Youth With Substance Use Disorders and Severe Mood Dysregulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-39577; 5K12DA000357-17 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-07-27 (Estimated); Results first posted 2022-04-18 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Substance Use Disorders; Bipolar Disorder; Mood Disorders
Keywords: youth; adolescent; young adult; substance use disorder; bipolar disorder; quetiapine; mood dysregulation
MeSH Terms: conditions — Substance-Related Disorders; Bipolar Disorder; Mood Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quetiapine (Experimental): Quetiapine
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Quetiapine — Participants will be randomly assigned Quetiapine and will be titrated to the maximum daily dose over three weeks and then enter a dose maintenance phase for weeks 4 through 8 of the study.
  Other Names: Seroquel
  Arms: Quetiapine
Other: Placebo — Participants will be randomly assigned to placebo and will be titrated to the maximum daily dose over three weeks and then enter a dose maintenance phase for weeks 4 through 8 of the study.
  Arms: Placebo

SUMMARY:
This study proposes to use quetiapine as an adjunct treatment to treatment as usual to improve both substance use disorder (SUD) and mood symptoms in youth with SUD and severe mood dysregulation (SMD). This is a randomized, double blind placebo controlled parallel design study. Youth with symptoms of mood dysregulation and active substance use that meets criteria for a SUD will be randomized to adjunct treatment with quetiapine or placebo. The investigators hypothesize that treatment with quetiapine will lead to a reduction in substance use, improvement in mood, and lead to greater engagement in outpatient treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 15 to 24
* Meet DSM-5 criteria for a substance use disorder
* Substance use ≥ 14 days of past 28 days (i.e. use ≥ 50% of days in the past 28 days)
* If subject in restricted setting/care (e.g. inpatient detox unit or residential treatment) for ≤ 2 weeks, then use ≥ 50% of days while outside of restricted setting (e.g. 7 days of substance use out of 14 days in unrestricted setting)
* Subjects need to have been in an unrestricted setting for at least 2 weeks prior to screening
* Meets DSM-5 criteria for bipolar disorder or disruptive mood dysregulation disorder or DSM IV criteria for mood disorder not otherwise specified
* Symptoms of SMD: Youth Self Report (YSR) or Adult Self Report (ASR) AAA ≥180
* Stable to be treated in outpatient level of care

Exclusion Criteria:

* Current methamphetamine use disorder
* Current unstable opioid use disorder (i.e. < 3 months on medication assisted treatment for an opioid use disorder)
* Pregnant or breastfeeding
* Placement in a restricted setting (e.g. detox or residential treatment) for ≥ 2 weeks out of past 28 days prior to screening visit, or placement in a restricted setting at anytime during study participation
* Unwilling or unable to use effective birth control
* Unwilling or unable to sign release of information for the treatment program providing behavioral treatment
* For participants >17 years-unable or unwilling to identify emergency contact

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Yule, M.D., Study Chair — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quetiapine | Placebo
Started | 13 | 11
Took One Dose of Study Medication | 11 | 10
Took One Week of Study Medication | 10 | 9
Completed | 7 | 6
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine | Placebo | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.2 (2.1) | 20.5 (1.8) | 20.8 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 9 | 6 | 15
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24
Beck Depression Inventory-II (BDI-II) [Mean (Standard Deviation); unit: Score on a scale] — The BDI-II assesses depressive symptomatology over the 2 weeks prior to administration. It is a 21-item scale with each question rated with a Likert rating scale from 0 to 3, and the total score representing a summation of all responses ranging from 0 to 63, with higher scores indicating greater impairment. Population: Data only available for participants who took at least one week of study medication.
  Score on a scale
    number analyzed (Participants) | 10 | 9 | 19
    (all) | 25 (9.5) | 25.9 (9) | 25.4 (9)
Young Mania Rating Scale [Mean (Standard Deviation); unit: Score on a scale] — The YMRS is composed of 11 items, each rated with a Likert rating scale. Each item is composed of 5 explicitly defined levels of severity. Severity ratings for 7 items are scored on a scale of 0 -4. The remaining 4 items are double weighted to account for poor cooperation of client when unwell and are scored on a scale of 0 - 8. Item ratings are sum to produce a total YMRS score between 0 -60. Higher scores on the YMRS indicate greater symptoms of mania. Population: Data only available for participants who took at least one week of study medication.
  Score on a scale
    number analyzed (Participants) | 10 | 9 | 19
    (all) | 18.8 (4.9) | 14.6 (5.4) | 16.9 (5.4)
Weiss Craving Scale [Mean (Standard Deviation); unit: Score on a scale] — The Weiss Craving Scale is a 3-item scale with each question rated with a Likert scale from 0 (no desire/likelihood of use) to 9 (strong desire/likelihood of use), and the total score representing the summation of all responses ranging from 0 to 27, with higher scores indicating more severe cravings. Population: Data only available for participants who took at least one week of study medication.
  Score on a scale
    number analyzed (Participants) | 10 | 9 | 19
    (all) | 17.1 (5.7) | 16.4 (6.3) | 16.8 (5.8)
Number of Participants with a Negative Urine Screen at Baseline [Number; unit: Participants] — Participants who took at least one week of study medication, completed at least one post-baseline urine toxicology screen, and whose drug of choice could be assessed with urine toxicology testing. Population: Data only available for participants who took at least one week of study medication, completed at least one post-baseline urine toxicology screen, and whose drug of choice could be assessed with urine toxicology testing.
  Participants
    number analyzed (Participants) | 8 | 7 | 15
    (all) | 1 | 2 | 3
Timeline Followback of Substance Use (TLFB) [Mean (Standard Deviation); unit: days] — The TLFB is used to quantify self-reported drug of choice use during the past month. Counts the number of days with substance use in the past 28 days. Population: Data only available for participants who took at least one week of study medication, and 28 days of information on timeline follow back for substance use after starting study medication.
  days
    number analyzed (Participants) | 8 | 8 | 16
    (all) | 19.5 (9.3) | 15.4 (8.2) | 17.4 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Timeline Followback of Substance Use (TLFB)
Description: The TLFB is used to quantify self-reported drug of choice use during the past month. Counts the number of days with substance use in the past 28 days.
Time Frame: baseline, 8 weeks
Population: Participants who completed at least one week of study medication and had 28 days-worth of past substance use data at baseline and study endpoint.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 8 | 8
Days | 2.3 (6.9) | 3.3 (6)

2. Primary Outcome: Change in Symptoms of Mania
Description: Symptoms of mania will be assessed using the Young Mania Rating Scale (YMRS). The YMRS consists of 11 items rated on a scale. Each item is composed of 5 explicitly defined levels of severity. Severity ratings for 7 items are scored on a scale of 0 -4. The remaining 4 items are double weighted to account for poor cooperation of client when unwell and are scored on a scale of 0 - 8. Item ratings are sum to produce a total YMRS score between 0 -60. Higher scores on the YMRS indicate greater symptoms of mania.
Time Frame: baseline, 8 weeks
Population: Participants who took at least one week of study medication and completed the YMRS at baseline and at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 10 | 8
score on a scale | -8.8 (8.1) | -0.4 (7.5)

3. Secondary Outcome: Change in the Number of Negative Urine Toxicology Specimens
Description: Urine toxicology specimens for the participant's drug of choice assessed as positive or negative. For each participant, the proportion of urine toxicology specimens that are negative over the course of the trial are calculated as the number of negative specimens divided by the total number of specimens collected from week 1 until study endpoint.
Time Frame: baseline, 8 weeks
Population: Participants who took at least one week of study medication, completed at least one post-baseline urine toxicology screen, and whose drug of choice could be assessed with urine toxicology testing.
Measure: Median (Inter-Quartile Range); unit: Proportion of Specimens
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 8 | 8
Proportion of Specimens | 0 [0 to 0.14] | 0 [0 to 0]

4. Secondary Outcome: Change in Craving for the Substance That the Participant Identifies as Most Problematic
Description: Craving will be measured by the Weiss Craving Scale. This scale consists of 3 items rated on a scale from 0 (no desire/likelihood of use) to 9 (strong desire/likelihood of use). The total Weiss Craving Scale score ranges from 0 to 27. Higher scores on the Weiss Craving Scale indicate greater cravings for a substance.
Time Frame: baseline, 8 weeks
Population: Participants who took at least one week of study medication and completed the Weiss Craving Scale at baseline and at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | -1.8 (4.5) | 0.4 (4.8)

5. Secondary Outcome: Change in Symptoms of Depression
Description: Symptoms of depression will be assessed using the Beck Depression Inventory II (BDI-II) scale. The BDI-II consists of 21 items rated on a scale from 0 (symptoms not present) to 3 (symptoms extremely severe). Total scores on the BDI-II range from 0 to 63. Higher scores indicate greater symptoms of depression.
Time Frame: baseline, 8 weeks
Population: Participants who took at least one week of study medication and completed the BDI-II at baseline and at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Quetiapine | Placebo
Number analyzed (Participants) | 10 | 9
score on a scale | -9.1 (13.5) | -6.2 (10.6)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Quetiapine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quetiapine (N=11) | Placebo (N=10)
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tootheache (Nervous system disorders) | 1 (1) | 0 (0)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 3 (3)
Burn on Skin (General disorders) | 0 (0) | 1 (2)
Chest Pain (Vascular disorders) | 1 (1) | 0 (0)
Nausea/Vomitting (Gastrointestinal disorders) | 3 (8) | 4 (5)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 5 (6)
Fatigue/Drowsiness/Sedation (General disorders) | 10 (24) | 4 (7)
Decreased Appetite (Gastrointestinal disorders) | 2 (4) | 1 (1)
Upset Stomach/Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Stomach Cramps (Gastrointestinal disorders) | 1 (3) | 0 (0)
Dizziness (General disorders) | 1 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal Yeast Infection (Infections and infestations) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Visual Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 5 (17)
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1)
Increased Appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
Increased General Anxiety (Psychiatric disorders) | 0 (0) | 1 (3)
Increased Thirst and Dry Mouth (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HSV Outbreak on Tailbone (Infections and infestations) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Sleep Paralysis (Psychiatric disorders) | 1 (1) | 0 (0)
Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/53/NCT02845453/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT02845453/ICF_002.pdf